CLINICAL TRIAL: NCT03677986
Title: Buprenorphine Treatment Engagement and Overdose Prevention in Opioid Users
Brief Title: Buprenorphine Treatment Engagement and Overdose Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00186156; R01CE003069-01 (NIH)
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-07

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants in this group will be referred to receive office-based buprenorphine treatment
- Video DOT+ (Experimental): Participants in this group will be referred to receive office-based buprenorphine treatment and will receive financial incentives for taking their daily buprenorphine dose.
  Interventions: Behavioral: Video DOT+

INTERVENTIONS:
Behavioral: Video DOT+ — Participants will receive financial incentives for recording and submitting videos of themselves taking their daily buprenorphine dose.
  Arms: Video DOT+

SUMMARY:
Office-based buprenorphine could be expanded to treat many of the opioid users who are not in treatment and who are at great risk for opioid overdose, but effective approaches are needed to help individuals with opioid use disorder initiate and remain in office-based buprenorphine treatment. Investigators propose to develop and pilot test a novel intervention that will combine video-based directly observed therapy and incentives to promote buprenorphine treatment engagement and adherence in out-of-treatment opioid users.

DETAILED DESCRIPTION:
The United States is experiencing an epidemic of opioid-related overdose deaths. Office-based buprenorphine treatment could expand access to treatment to the many opioid users who are not in treatment and who are at great risk for opioid overdose. However, office-based buprenorphine has two limitations that Investigators will address in this application: 1) Patients prescribed buprenorphine by office-based providers can divert the buprenorphine for illicit use. 2) Many people in need of buprenorphine treatment do not initiate and remain in office-based buprenorphine treatment. Investigators will use Video Directly Observed Therapy (DOT) and incentives to enhance office-based buprenorphine treatment. Video DOT is an innovative, mobile health platform that patients can use to record and submit videos of patients taking medication that are then viewable on a secure, web portal for providers to confirm medication adherence. Video DOT could facilitate adherence to buprenorphine treatment and safeguard against diversion. The addition of incentives could engage out-of-treatment opioid users into treatment and increase treatment retention. Incentive interventions, which provide incentives to patients meeting therapeutic goals, have been highly effective in promoting a wide range of health behaviors and have firm theoretical and empirical foundations. Incentive interventions can promote treatment engagement in individuals with substance use disorders, including out-of-treatment opioid users. Investigators propose to develop and pilot test a novel combination of Video DOT and incentives to promote buprenorphine treatment engagement and adherence in out-of-treatment opioid users. The Video DOT+ intervention will provide an incentive for linking to buprenorphine treatment and facilitate retention in treatment by providing incentives for maintaining daily buprenorphine use as verified by the Video DOT system. The incentives will be integrated into the Video DOT platform and delivered remotely to reloadable credit cards to allow for the entire intervention to be delivered via mobile technology and to facilitate easy dissemination of the Video DOT+ system. A randomized pilot study is planned over 3 years. Out-of-treatment opioid users (N=64) will be referred to buprenorphine treatment and randomly assigned to a Usual Care (Control) group or Video DOT+ group. Video DOT+ participants will receive the Video DOT+ intervention being developed and evaluated in this project. Investigators will assess participants every 4 weeks throughout a 24-week intervention period and at 12 weeks after the intervention ends. The primary outcome measure will be buprenorphine treatment adherence during the 24-week intervention. Secondary measures will include buprenorphine treatment engagement (linkage and retention), opioid use, risk of opioid overdose, and post-intervention effects. The project will allow for the development and preliminary evaluation of a novel intervention to promote buprenorphine treatment engagement and adherence in out-of-treatment opioid users. Ultimately, Investigators would like to develop and disseminate an effective and scalable intervention that can enhance office-based buprenorphine treatment and thereby combat the opioid overdose epidemic.

ELIGIBILITY:
Inclusion Criteria:

* opioid use disorder

Exclusion Criteria:

* current suicidal/homicidal ideation
* severe psychiatric disorder

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, Ph.D., Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Center for Learning and Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toegel F, Novak MD, Rodewald AM, Leoutsakos JM, Silverman K, Holtyn AF. Technology-assisted opioid education for out-of-treatment adults with opioid use disorder. Psychol Addict Behav. 2022 Aug;36(5):555-564. doi: 10.1037/adb0000769. Epub 2021 Jul 29. PMID 34323526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via community agencies that served the target population and a referral system in which study participants were paid for successfully referring others to the study. Interested individuals completed a brief phone interview. Potentially eligible participants were invited for a full in-person interview.
Groups:
- Video DOT+: Participants in this group will be referred to receive office-based buprenorphine treatment and will receive financial incentives for taking their daily buprenorphine dose.
  Video Directly Observed Therapy (DOT)+: Participants will receive financial incentives for recording and submitting videos of themselves taking their daily buprenorphine dose.
Period: Overall Study
Arm/Group | Usual Care | Video DOT+
Started | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Video DOT+ | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (8.9) | 44.6 (11.4) | 46.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 11 | 28
  White | 1 | 10 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 21 | 41
Self-reported methadone use [Count of Participants; unit: Participants] — Participants reporting methadone use.
  Participants | 6 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Buprenorphine Treatment Adherence
Description: This will be assessed by the percentage of buprenorphine-positive urine samples during the 24-week intervention.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: percentage of urine samples
Arm/Group | Usual Care | Video DOT+
Number analyzed (Participants) | 20 | 21
percentage of urine samples | 19.7 (4.0) | 16.1 (3.7)
Statistical Analysis 1: Comparison: Usual Care vs Video DOT+; Test type: Superiority; p = 0.914, GEE; Odds Ratio (OR) = 0.92, 95% CI 2-sided [.21 to 4.14]

2. Secondary Outcome: Linkage to Treatment
Description: This will be assessed by the percentage of participants who get linked to buprenorphine treatment during the 24-week intervention
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: To monitor adverse events, all staff members are instructed on the need to report to an investigator any indication that an adverse event has occurred. When the staff members and investigators learn of an adverse event, they will investigate until they have determined as many of the relevant details of the adverse event as possible. Also, participants will be asked about all categories of adverse events at each routine assessment visit conducted throughout the studies.
Arm/Group | Usual Care | Video DOT+
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT03677986/Prot_SAP_000.pdf